CLINICAL TRIAL: NCT02955641
Title: Efficacy and Necessity of Anti-inflammatory Drops After Laser Peripheral Iridotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-16-3197-AL-CTIL
Record Dates: First submitted 2016-09-05; First posted 2016-11-04 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma, Closed-Angle; Glaucoma, Narrow-Angle; Glaucoma, Angle-Closure
Keywords: Laser peripheral iridotomy; topical anti-inflammatory drops
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — nepafenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- NSAIDs-Placebo (Active Comparator): Will receive Nepafenac 0.1%in the first eye, and Hydroxyethylcellulose 0.19% in the second eye
  Interventions: Drug: Nepafenac 0.1%; Drug: Hydroxyethylcellulose 0.19%
- Placebo-NSAIDs (Active Comparator): Will receive Hydroxyethylcellulose 0.19% in the first eye, and Nepafenac 0.1%in the second eye
  Interventions: Drug: Nepafenac 0.1%; Drug: Hydroxyethylcellulose 0.19%
- Steroid-Placebo (Active Comparator): Will receive Dexamethasone Disodium Phosphate 0.1% in the first eye, and Hydroxyethylcellulose 0.19% in the second eye
  Interventions: Drug: Dexamethasone Disodium Phosphate 0.1%; Drug: Hydroxyethylcellulose 0.19%
- Placebo-Steroids (Active Comparator): Will receive Hydroxyethylcellulose 0.19%in the first eye, and Dexamethasone Disodium Phosphate 0.1%in the second eye
  Interventions: Drug: Dexamethasone Disodium Phosphate 0.1%; Drug: Hydroxyethylcellulose 0.19%

INTERVENTIONS:
Drug: Dexamethasone Disodium Phosphate 0.1% — four drops a day for four days after LPI treatment
  Other Names: Sterodex
  Arms: Placebo-Steroids; Steroid-Placebo
Drug: Nepafenac 0.1% — four drops a day for four days after LPI treatment
  Other Names: Nevanac
  Arms: NSAIDs-Placebo; Placebo-NSAIDs
Drug: Hydroxyethylcellulose 0.19% — four drops a day for four days after LPI treatment
  Other Names: Lyteers ophthalmic solution

SUMMARY:
The purpose of this study is to evaluate the efficacy and need for prescribing anti-inflammatory topical drops to patients undergoing laser peripheral iridotomy.

DETAILED DESCRIPTION:
Primary closed angle glaucoma is responsible to almost half glaucoma related blindness around the world. Laser peripheral iridotomy (LPI) is a common and simple treatment used for both treatment and prevention of acute angle closure event.

Anti-inflammatory drops are commonly prescribed to patients undergoing LPI in order to prevent or reduce post-treatment discomfort. However, to date, there are no specific guidelines for post LPI anti-inflammatory treatment, nor sufficient clinical evidence regarding the efficacy of such treatment.

In the current study, the investigators aim to evaluate the effect of topical steroids and non-steroidal anti-inflammatory drugs (NSAIDs) on post LPI symptoms and inflammation markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary narrow/closed angle by gonioscopy
* Able to give consent
* Ability to attend follow-up visits

Exclusion Criteria:

* Corneal disease preventing sufficient evaluation of the angle
* Secondary closed angle (e.g. uveitis related)
* Pregnant women
* Previous eye surgery other than laser refractive correction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Pain score | At four days post LPI treatment
  Using VAS pain scale
Symptoms score | At four days post LPI treatment
  Using a modified questionnaire based on the ocular surface disease index.

SECONDARY OUTCOMES:
Grading of cells in the anterior chamber | At four days post LPI treatment
  Assessed by counting the number of cells in the anterior chamber and applying the SUN working group grading scheme for anterior chamber cells
Patency of LPI by visualisation | up to 30 days post LPI treatment
  Assessed on slit-lamp examination using transilumination and visualising the site of LPI treatment for the presence (patent) or obsence (closed) of transilumination defect
Grading of flare in anterior chamber | At four days post LPI treatment
  Assessed by counting the number of cells in the anterior chamber and applying the SUN working group grading scheme for anterior chamber flare

CONTACTS AND LOCATIONS:
Overall Officials: Ari Leshno, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: Undecided